CLINICAL TRIAL: NCT04564612
Title: An Open-Label, Pharmacokinetic Study to Evaluate the Pharmacokinetics and Relative Bioavailability of BIIB091 Formulations and to Assess the Impact of Food, a Proton Pump Inhibitor and CYP3A4 Inhibitor on BIIB091 Exposure Using the Selected Formulation in Healthy Subjects
Brief Title: Study of BIIB091 Formulations in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 257HV105; 2020-000682-16 (EudraCT Number)
Record Dates: First submitted 2020-09-21; First posted 2020-09-25 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — BIIB091; Rabeprazole; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1 (Experimental): Participants will receive single oral dose of BIIB091 on Day 1 of each study period, in fasted state, for up to 5 periods. There will be a minimum 7-day washout between Day 1 of each study period.
  Interventions: Drug: BIIB091
- Part 1B (Experimental): Participants will be randomized to receive single oral or 2 oral doses for divided daily doses of BIIB091 on Day 1 of Period 1, in fasted state or single oral dose of BIIB091 on Day 1 of Period 1, in fed state. Participants will receive single oral dose of BIIB091 on Day 1 of Period 2, in fasted state. Participants will receive single or two divided oral dose(s) of BIIB091 on Day 1 of Periods 3 and 4, in fasted or fed state. There will be a minimum 7-day washout between Day 1 of each study period.
  Interventions: Drug: BIIB091
- Part 2 (Experimental): Participants will receive single oral dose of BIIB091 on Day (D) 1 of Period (P) 1 in fasted/fed state; then itraconazole 100 milligram (mg) capsules (cap), orally, twice daily (BID) for 1 day (D -4) of P2, in fed state; then itraconazole 100 mg cap, orally, once daily (QD) for 2 days (D -3, -2) of P2, in fed state; then itraconazole 100 mg cap, orally, QD for 1 day (D -1) of P2, in fasted/fed state; then combination of itraconazole 100 mg cap, orally and BIIB091, orally on 5th day (D 1) of P2, in fasted/fed state; then itraconazole 100 mg cap, orally on 6th day (D 2) of P2, in fed state; then rabeprazole 20 mg tablets (tab), orally, BID for 3 days (D -3, -2, and -1) of P3 in fed state; then combination of rabeprazole 20 mg tab, orally and BIIB091, orally, on 4th day (D 1) of P3 in fasted/fed state. Minimum 7-day washout between dose of BIIB091 in P1 and 1st dose of itraconazole in P2; minimum 10-day washout between final dose of itraconazole in P2 and 1st dose of rabeprazole in P3.
  Interventions: Drug: BIIB091; Drug: Rabeprazole; Drug: Itraconazole
- Part 3 (Experimental): Participants will receive BIIB091, orally, QD or BID for at least 7 days in fasted or fed state.
  Interventions: Drug: BIIB091

INTERVENTIONS:
Drug: BIIB091 — Administered as specified in the treatment arm
Drug: Rabeprazole — Administered as specified in the treatment arm
  Arms: Part 2
Drug: Itraconazole — Administered as specified in the treatment arm
  Arms: Part 2

SUMMARY:
The primary objectives of this study are: to evaluate the pharmacokinetic (PK) profiles of BIIB091 modified release (MR) formulations in healthy participants after single dose administration in the fasted state (Part 1); to evaluate the PK profile of the BIIB091 immediate release (IR) tablet formulation in healthy participants after single dose administration (Part 1B); to determine the relative bioavailability of single doses of the selected BIIB091 regimen in healthy participants taking a proton pump inhibitor (PPI) compared to healthy participants not taking a PPI, to determine the relative bioavailability of single doses of the selected BIIB091 regimen in healthy participants taking a cytochrome P450 (CYP)3A4 inhibitor compared to healthy participants not taking a CYP3A4 inhibitor (Part 2); to evaluate the PK of the selected BIIB091 regimen in healthy participants after multiple dose administration (Part 3).

The secondary objectives of this study are: to determine the relative bioavailability of a single dose of the BIIB091 MR formulations compared to that of the IR drug in capsule (DiC) reference formulation in healthy participants in the fasted state, to assess the safety and tolerability of single doses of BIIB091 when administered as MR formulations in healthy participants in the fasted state (Part 1); to determine the PK of a single dose of the BIIB091 IR tablet formulation in the fed and fasted state in healthy participants, to evaluate the PK profiles of the BIIB091 IR tablet formulation in healthy participants after administration of divided total daily doses over a 24 hour period in the fasted or fed state, to determine the relative bioavailability of a single dose or divided dose of the BIIB091 IR tablet formulation compared to that of the IR DiC reference formulation in healthy participants in the fasted state, to determine the PK of a single or divided dose of the BIIB091 IR tablet formulation administered with an alternative meal composition in healthy participants, to assess the safety and tolerability of a single or divided dose of BIIB091 when administered as the IR tablet formulation and IR DiC reference formulation in healthy participants in fed or fasted state (Part 1B); to confirm the PK profiles of the selected BIIB091 regimen in healthy participants after single dose administration, and to establish a reference exposure for the assessment of drug interaction, to assess the safety and tolerability of single doses of BIIB091 when administered as the selected BIIB091 regimen in healthy participants taking a PPI, to assess the safety and tolerability of single doses of BIIB091 when administered as the selected BIIB091 regimen in healthy participants taking a CYP3A4 inhibitor (Part 2); to assess the safety and tolerability of multiple doses of BIIB091 when administered as the selected BIIB091 regimen in healthy participants (Part 3).

ELIGIBILITY:
Key Inclusion Criteria:

* Have a body mass index (BMI) between 18.0 and 30.0 kilograms per meter square (kg/m^2), inclusive, and a body weight of at least 50 kilogram (kg), as measured at screening.
* Must be in good health as determined by the Investigator, based on medical history and screening evaluations.
* A negative test for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) according to local guidelines, at screening and admission or prior to admission.

Key Exclusion Criteria:

* History of any clinically significant cardiac, endocrine, GI, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, or renal disease, or other major disease, as determined by the Investigator.
* Clinically significant 12-lead ECG abnormalities at screening and prior to first dose, including confirmed demonstration of QT interval corrected for heart rate using Fridericia's formula (QTcF) >450 milliseconds (msec), QRS >120 msec, PR >220 msec, or heart rate <50 beats per minute (bpm) based on the average of triplicate measurements, early repolarization, or any other clinically significant 12-lead ECG abnormalities as determined by the Investigator.
* History of torsades de pointes or additional risk factors for torsades de pointes (e.g. heart failure, hypokalemia, family history of long QT syndrome, or any medications known to prolong QT interval administered within 5.5 half-lives prior to screening), in the opinion of the Investigator.
* Receipt of any vaccination within 30 days prior to screening, or plans to receive the same any time from screening through to 30 days after the last study visit. However, non-live coronavirus disease 2019 (COVID-19) vaccination will be permitted 21 days or more prior to the first dose of BIIB091, as per local regulation and Investigator discretion.
* Evidence of current SARS-CoV-2 infection within the past 4 weeks at screening, between screening and admission, or at admission, including but not limited to any of the following symptoms: fever (temperature more than {>} 37.5 degree Celsius {°C}), new and persistent cough, breathlessness, or loss of taste or smell as per the judgement of the Investigator.
* Contact with an individual with COVID-19 infection in the past 14 days at screening, between screening and admission, or at admission.
* Presence or history of chronic, recurrent, or serious infection, as determined by the Investigator, within 90 days prior to screening or between screening and admission.
* Clinically significant abnormal laboratory test values, as determined by the Investigator, at screening.
* Current enrollment or plan to enroll in any other drug, biological, device, or clinical study, or treatment with an investigational drug or approved therapy for investigational use within 90 days prior to Day 1, or 5 half-lives of the drug or therapy, whichever is longer.
* Use of CYP3A4 inducers or inhibitors (including hormonal contraceptives as applicable) within 14 days before the first dose of study medication. Use of organic anion transporting polypeptide 1 (OATP1) B1 and B3 substrates in the 14 days before first dose of study medication.
* Chronic use of immunosuppressive or immunomodulatory drugs within 6 months prior to admission. (Recent acute use of immunosuppressants should be discussed with Sponsor.)
* Consumption of any product containing grapefruit, pomelos, or Seville oranges within 14 days of admission and an unwillingness to refrain from such products during study participation.
* Participants who have previously been enrolled in this study.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2022-09-07 (Actual); Study Completion 2022-09-07 (Actual)

PRIMARY OUTCOMES:
Parts 1 and 1B: Time Prior to the First Measurable Concentration (Tlag) of BIIB091 | Part 1: Up to Day 4; Part 1B: Up to Day 5
Parts 1, 1B and 3: Time of Maximum Observed Concentration (Tmax) of BIIB091 | Part 1: Up to Day 4; Part 1B: Up to Day 5; Part 3: Up to Day 14
Parts 1, 1B and 3: Maximum Observed Concentration (Cmax) of BIIB091 | Part 1: Up to Day 4; Part 1B: Up to Day 5; Part 3: Up to Day 14
Parts 1 and 1B: Plasma Concentration at 12 Hours (C12h) of BIIB091 | Parts 1 and 1B: 12 hours post-dose (Day 1)
Parts 1 and 1B: Plasma Concentration at 24 Hours (C24h) of BIIB091 | Parts 1 and 1B: 24 hours post-dose (Day 2)
Parts 1 and 1B: Area Under the Curve from Time 0 to 12 Hours Post-Dose [AUC(0-12h)] of BIIB091 | Parts 1 and 1B: Up to 12 hours post-dose (Day 1)
Parts 1 and 1B: Area Under the Curve from Time 0 to 24 Hours Post-Dose [AUC(0-24h)] of BIIB091 | Parts 1 and 1B: Up to 24 hours post-dose (Day 2)
Parts 1 and 1B: Area Under the Curve from Time 0 to the Time of Last Measurable Concentration [AUC(0-last)] of BIIB091 | Part 1: Up to Day 4; Part 1B: Up to Day 5
Parts 1, 1B and 3: Area Under the Curve from Time 0 Extrapolated to Infinity [AUC(0-inf)] of BIIB091 | Part 1: Post-dose at multiple time points up to Day 4; Part 1B: Post-dose at multiple time points up to Day 5; Part 3: Post-dose at multiple time points up to Day 14
Parts 1 and 1B: Area Under the Curve from Time of the Last Measurable Concentration to Infinity as a Percentage of the Area Under the Curve Extrapolated to Infinity (AUC%extrap) of BIIB091 | Part 1: Up to Day 4; Part 1B: Up to Day 5
Parts 1, 1B and 3: Terminal Elimination Half-Life (T1/2) of BIIB091 | Part 1: Up to Day 4; Part 1B: Up to Day 5; Part 3: Up to Day 14
Parts 1, 1B and 3: First Order Rate Constant Associated with the Terminal (Log-Linear) Portion of the Curve (Lambda-z) of BIIB091 | Part 1: Up to Day 4; Part 1B: Up to Day 5; Part 3: Up to Day 14
Parts 1 and 1B: Total Body Clearance of BIIB091 Calculated After a Single Extravascular Administration Where Fraction of Dose Bioavailable (F) is Unknown (CL/F) | Part 1: Up to Day 4; Part 1B: Up to Day 5
Parts 1 and 1B: Apparent Volume of Distribution of BIIB091 Based on the Terminal Phase Calculated Using AUC(0-inf) After a Single Extravascular Administration Where F is Unknown (Vd/F) | Part 1: Up to Day 4; Part 1B: Up to Day 5
Part 2: Relative Bioavailability of BIIB091 Based on Cmax (Frel Cmax) of BIIB091 Dosed With and Without Proton Pump Inhibitor (PPI) | Part 2: Up to Day 5
Part 2: Relative Bioavailability of BIIB091 Based on AUC(0-last) [Frel AUC(0-last)] of BIIB091 Dosed With and Without PPI | Part 2: Up to Day 5
Part 2: Relative Bioavailability of BIIB091 Based on AUC(0-inf) [Frel AUC(0-inf)] of BIIB091 Dosed With and Without PPI | Part 2: Up to Day 5
Part 2: Frel Cmax of BIIB091 Dosed With and Without Cytochrome P450 (CYP) 3A4 Inhibitor | Part 2: Up to Day 5
Part 2: Frel AUC(0-last) of BIIB091 Dosed With and Without CYP3A4 Inhibitor | Part 2: Up to Day 5
Part 2: Frel AUC(0-inf) of BIIB091 Dosed With and Without CYP3A4 Inhibitor | Part 2: Up to Day 5
Part 3: Concentration at the End of the Dosing Interval (Ctrough) of BIIB091 | Part 3: Up to Day 14
Part 3: Area Under Curve Observed at the End of the Dosing Interval (AUCtau) of BIIB091 | Part 3: Up to Day 14
Part 3: Plasma Concentration Observed at the End of the Dosing Interval (Ctau) of BIIB091 | Part 3: Up to Day 14
Part 3: Minimum Observed Concentration (Cmin) of BIIB091 | Part 3: Up to Day 14
Part 3: Average Concentration (Cave) of BIIB091 | Part 3: Up to Day 14
Part 3: Peak to Trough Fluctuation | Part 3: Up to Day 14
  The formula used will be (Cmax-Cmin)/average concentration (Cavg) × 100.
Part 3: Accumulation Ratio Based on Cmax/Cmax Single Dose (AR Cmax) | Part 3: Up to Day 14
Part 3: Accumulation Ratio Based on AUCtau/AUCtau Single Dose (AR AUCtau) | Part 3: Up to Day 14
Part 3: Total Body Clearance Calculated Using AUCtau After Repeated Extravascular Administration Where F is Unknown (CL/Ftau) | Part 3: Up to Day 14
Part 3: Apparent Volume of Distribution Based on the Terminal Phase Calculated Using AUCtau After Extravascular Administration Where F is Unknown (Vd/Ftau) | Part 3: Up to Day 14

SECONDARY OUTCOMES:
Parts 1 and 1B: Frel Cmax of BIIB091 | Part 1: Up to Day 4; Part 1B: Up to Day 5
  Parameter will be evaluated for the fed versus (vs) fasted comparison and the alternative meal composition comparison.
Parts 1 and 1B: Frel AUC(0-last) of BIIB091 | Part 1: Up to Day 4; Part 1B: Up to Day 5
  Parameter will be evaluated for the fed vs fasted comparison and the alternative meal composition comparison.
Parts 1 and 1B: Frel AUC(0-inf) of BIIB091 | Part 1: Up to Day 4; Part 1B: Up to Day 5
  Parameter will be evaluated for the fed vs fasted comparison and the alternative meal composition comparison.
Parts 1, 1B, 2 and 3: Number of Participants with Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | From Signing of Informed Consent Form (ICF) Until Follow-up Phone Call (Parts 1 and 1B: Up to 15 weeks; Part 2: Up to 10 weeks; Part 3: Up to 7 weeks)
  An adverse event (AE) is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An SAE is any untoward medical occurrence that at any dose results in death, places the participant at immediate risk of death, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, results in a congenital anomaly/birth defect or is a medically important event.
Parts 1, 1B, 2 and 3: Number of Participants with Electrocardiogram (ECG) Abnormalities as Assessed by 12-Lead ECG Measurements | Part 1: Up to Day 4; Parts 1B and 2: Up to Day 5; Part 3: Up to Day 14
Parts 1B and 2: Time Prior to the First Measurable Concentration (Tlag) of BIIB091 | Parts 1B and 2: Up to Day 5
  Parameter will be evaluated for the fed vs fasted comparison and the alternative meal composition comparison in Part 1B.
Parts 1B and 2: Time of Maximum Observed Concentration (Tmax) of BIIB091 | Parts 1B and 2: Up to Day 5
  Parameter will be evaluated for the fed vs fasted comparison and the alternative meal composition comparison in Part 1B.
Parts 1B and 2: Maximum Observed Concentration (Cmax) of BIIB091 | Parts 1B and 2: Up to Day 5
  Parameter will be evaluated for the fed vs fasted comparison and the alternative meal composition comparison in Part 1B.
Parts 1B and 2: Plasma Concentration at 12 Hours (C12h) of BIIB091 | Parts 1B and 2: 12 hours post-dose (Day 1)
  Parameter will be evaluated for the fed vs fasted comparison and the alternative meal composition comparison in Part 1B.
Parts 1B and 2: Plasma Concentration at 24 Hours (C24h) of BIIB091 | Parts 1B and 2: 24 hours post-dose (Day 2)
  Parameter will be evaluated for the fed vs fasted comparison and the alternative meal composition comparison in Part 1B.
Parts 1B and 2: Area Under the Curve from Time 0 to 12 Hours Post-Dose [AUC(0-12h)] of BIIB091 | Parts 1B and 2: Up to 12 hours post-dose (Day 1)
  Parameter will be evaluated for the fed vs fasted comparison and the alternative meal composition comparison in Part 1B.
Parts 1B and 2: Area Under the Curve from Time 0 to 24 Hours Post-Dose [AUC(0-24h)] of BIIB091 | Parts 1B and 2: Up to 24 hours post-dose (Day 2)
  Parameter will be evaluated for the fed vs fasted comparison and the alternative meal composition comparison in Part 1B.
Parts 1B and 2: Area Under the Curve from Time 0 to the Time of Last Measurable Concentration [AUC(0-last)] of BIIB091 | Parts 1B and 2: Up to Day 5
  Parameter will be evaluated for the fed vs fasted comparison and the alternative meal composition comparison in Part 1B.
Parts 1B and 2: Area Under the Curve from Time 0 Extrapolated to Infinity [AUC(0-inf)] of BIIB091 | Parts 1B and 2: Post-dose at multiple time points up to Day 5
  Parameter will be evaluated for the fed vs fasted comparison and the alternative meal composition comparison in Part 1B.
Parts 1B and 2: Area Under the Curve from Time of the Last Measurable Concentration to Infinity as a Percentage of the Area Under the Curve Extrapolated to Infinity (AUC%extrap) of BIIB091 | Parts 1B and 2: Up to Day 5
  Parameter will be evaluated for the fed vs fasted comparison and the alternative meal composition comparison in Part 1B.
Parts 1B and 2: Terminal Elimination Half-Life (T1/2) of BIIB091 | Parts 1B and 2: Up to Day 5
  Parameter will be evaluated for the fed vs fasted comparison and the alternative meal composition comparison in Part 1B.
Parts 1B and 2: First Order Rate Constant Associated with the Terminal (Log-Linear) Portion of the Curve (Lambda-z) of BIIB091 | Parts 1B and 2: Up to Day 5
  Parameter will be evaluated for the fed vs fasted comparison and the alternative meal composition comparison in Part 1B.
Parts 1B and 2: Total Body Clearance of BIIB091 Calculated After a Single Extravascular Administration Where Fraction of Dose Bioavailable (F) is Unknown (CL/F) | Parts 1B and 2: Up to Day 5
  Parameter will be evaluated for the fed vs fasted comparison and the alternative meal composition comparison in Part 1B.
Parts 1B and 2: Apparent Volume of Distribution of BIIB091 Based on the Terminal Phase Calculated Using AUC(0-inf) After a Single Extravascular Administration Where F is Unknown (Vd/F) | Parts 1B and 2: Up to Day 5
  Parameter will be evaluated for the fed vs fasted comparison and the alternative meal composition comparison in Part 1B.
Part 1B: Relative Bioavailability of BIIB091 Based on AUC(0-24h) [Frel AUC(0-24h)] | Part 1B: Up to Day 5

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Research Site, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/